CLINICAL TRIAL: NCT00773487
Title: Influence of Diesel Exhaust Particles (DEP) With and Without Organic Compounds on the Allergic Inflammation in Asthmatic Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fraunhofer-Institute of Toxicology and Experimental Medicine (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Prof. Dr. Norbert Krug, Fraunhofer ITEM
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 08/06 DEP-SFB
Record Dates: First submitted 2008-10-14; First posted 2008-10-16 (Estimated); Last update posted 2009-07-28 (Estimated); Status verified 2009-07

CONDITIONS: Asthma
Keywords: Asthma GINA 1; Mild intermittant asthma
MeSH Terms: conditions — Asthma

INTERVENTIONS:
Other: Bonchoscopy — Segmental instillation of allergen/Diesel particles; bronchoalveolar lavage

SUMMARY:
The primary objective of this study is to elucidate the effects of Diesel particles on the allergic inflammation in the airways of asthmatic patients.

DETAILED DESCRIPTION:
A first bronchoscopy will be performed with a baseline bronchoalveolar lavage (BAL) and epithelial brushes followed by a segmental instillation of allergen (grass mix or house dust mite) alone, in combination with Diesel particles, further in combination with Diesel particles without organic compounds and saline as control into four different lung segments. After 24 hours, during a second bronchoscopy, BAL samples will be collected in these challenged segments in order to obtain cells and lavage fluid for cell biological and immunological analysis.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give written informed consent
* Physician diagnosis of mild intermittent or mild persistent asthma according to GINA guidelines {Bateman, 2008 34 /id}
* Age 18-55 years
* Nonsmokers with a history of less than 1 packyear having been nonsmokers for at least the last five years
* FEV1 >= 80% of predicted, FEV1/FVC >= 70 %
* Positive skin prick test for grass mix or D. pteronyssinus at or within 12 months prior to the screening visit
* Positive response to inhaled methacholine (<= 8mg/ml)
* Positive response to an incremental inhaled allergen challenge with house dust mite allergen or grass pollen allergen
* Available to complete all study measurements

Women will be considered for inclusion if they are:

* Not pregnant, as confirmed by pregnancy test, and not nursing
* Of non-child bearing potential (i.e. physiologically incapable of becoming pregnant, including any female who is pre-menarchial or post-menopausal, with documented proof of hysterectomy or tubal ligation, or meet clinical criteria for menopause and has been amenorrhoeic for more than 1 year prior to the screening visit)
* Of childbearing potential and using a highly effective method of contraception during the entire study (vasectomised partner, sexual abstinence - the lifestyle of the female should be such that there is complete abstinence from intercourse from two weeks prior to the study until at least 72 hours after the end of the study -, implants, injectables, combined oral contraceptives, hormonal IUDs)

Exclusion Criteria:

* History of upper or lower respiratory tract infection four weeks prior to the informed consent visit
* Past or present disease, which as judged by the investigator, may affect the outcome of this study. These diseases include, but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease, hematological disease, neurological disease, psychiatric disease, endocrine disease, infectious disease, inflammatory disease, or pulmonary disease (including but not confined to chronic bronchitis, emphysema, tuberculosis, bronchiectasis or cystic fibrosis).
* Clinically significant pathological findings in safety laboratory tests
* Regular intake of any medication other than short acting inhaled beta agonists, paracetamol for pain relief, birth control medication, hormonal replacement therapy, dietary and vitamin supplements
* Specific Immunotherapy (SIT) within two years prior to the study
* Use of anti-inflammatory medication including systemic or inhaled corticosteroid within the last four weeks
* Any history of life-threatening asthma, defined as an asthma episode that required intubation and/or was associated with hypercapnea, respiratory arrest or hypoxic seizures.
* Suspected hypersensitivity to any ingredients of the medication in line with bronchoscopy (bronchodilators, sedatives and local anesthetics)
* Conditions or factors, which would make the subject unlikely to be able to undergo bronchoscopy or incremental allergen challenge
* History of drug or alcohol abuse
* Suspected inability to understand the protocol requirements, instructions and study-related restrictions, the nature, scope, and possible consequences of the study.
* Participation in a clinical trial 30 days prior to enrolment
* Segmental allergen challenge 3 months prior to treatment
* Risk of non-compliance with study procedures

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
difference of the total number of eosinophils resulting in the comparison of allergic versus allergic inflammation in combination with Diesel particles with and without the organic fraction. | 24 post allergen challenge

CONTACTS AND LOCATIONS:
Overall Officials: Norber Krug, MD, Principal Investigator — Fraunhofer ITEM
Locations (1):
- Fraunhofer ITEM, Hanover, Lower Saxony, Germany